CLINICAL TRIAL: NCT01379131
Title: MI as the First Manifestation of Coronary Heart Disease: Distribution of Previous Cardiovascular Disease, Cardiovascular Risk Factors and Chest Pain in First MI
Brief Title: Previous Cardiovascular Disease, Cardiovascular Risk Factors and Chest Pain in First Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Emily Herrett, Dr, London School of Hygiene and Tropical Medicine
Other Study IDs: CALIBER 09-07b; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: Manifestation; Coronary Heart Disease; Myocardial infarction; Angina pectoris; Unheralded; General Practice Research Database; Myocardial Ischaemia National Audit Project; CALIBER
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Angina Pectoris

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GPRD patients: All patients included in "up to standard" GPRD practices that agreed to the linkage with the MINAP database are included in this cohort.

SUMMARY:
Some myocardial infarctions (MI) occur as the first manifestation of atherosclerotic disease. Such MIs are important because of the high likelihood of missed opportunities for prevention. A recent analysis using CALIBER data estimated this proportion at 60%.

Further to this research, another level of complexity can be added to improve our understanding of these MIs. This is the concept of a completely 'unanticipated' MI, which can be defined as: MI occurring as the first manifestation of atherosclerotic disease and without any traditional cardiovascular risk factors and without any prior chest pain. Such 'unanticipated' MIs cannot be foreseen by the medical profession and their frequency in the population is unknown.

Therefore the aim of this study is to describe the distribution of previously diagnosed cardiovascular disease, cardiovascular risk factors and chest pain in patients with first MI. This will provide an estimate of the number of 'unanticipated' MIs and of the levels of risk factors in unheralded, compared to heralded MI.

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

Using data from GPRD, MINAP, ONS mortality data and Hospital Episode Statistics (HES), this study will identify patients with a first MI (STEMI and non-STEMI). Information from in-patient hospital visits, general practice data and self-reported data in MINAP, this study will allow the quantification of the level and timing of cardiovascular disease before first MI. It will also measure the levels of cardiovascular risk factors and chest pain occurring before MI.

ELIGIBILITY:
Inclusion Criteria:

* Patients in GPRD practices which are deemed "up to standard" by GPRD criteria will be included if their practice agreed to be linked to the MINAP dataset.
* Age over 18.

Exclusion Criteria:

* Patients will be excluded after experiencing their first MI.
* Patients will be excluded if they do not fulfil one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients registered at those GPRD practices that agreed to the linkage with the MINAP database, and whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of all UK practices, and 98% of people in the UK are registered with a GP. Therefore the GPRD should be a representative sample of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
First myocardial infarction (MI) | Average time frame: up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Herrett, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom